CLINICAL TRIAL: NCT04842994
Title: Phase III, Assessor Blinded, Randomised Controlled Trial of Use of Intraoperative Neuromonitoring (IONM) in Thyroid Cancer Surgery(ACTION)
Brief Title: Trial on Intraoperative Neuromonitoring (IONM) in Thyroid Cancer Surgery.
Acronym: ACTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Gouri Pantvaidya, Professor and Consultant Surgeon Department of Head & Neck Surgery, Tata Memorial Centre Secretary, Data Safety Monitoring Unit, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3223
Record Dates: First submitted 2020-10-06; First posted 2021-04-13 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Malignant Neoplasm of Thyroid Gland
Keywords: Thyroid cancer; Intraoperative neuromonitoring; Recurrent laryngeal nerve palsy; randomised trial; acoustic analysis
MeSH Terms: conditions — Thyroid Neoplasms; Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IONM arm (Experimental): Intra operative nerve monitoring (IONM) is a technique of monitoring the RLN during surgery, to help identification and safe guarding of the nerve during total thyroidectomy as well as central compartment clearance (CCC). This is a well established technique with many centers in the world routinely using monitoring during surgery.
  Interventions: Device: IONM tube
- Visual Identification arm (No Intervention): Patients randomized to this arm will undergo total thyroidectomy as per standard procedures with visual identification of the RLNs

INTERVENTIONS:
Device: IONM tube — The standardized technique of IONM-RLNs (bilaterally) will be used, including indirect vagal response evaluation at the beginning and also at the end of surgery according to the recommendations formulated by the International Intraoperative Neural Monitoring Study Group (INMSG) (Randolph GW, Dralle H. 2011).
  Arms: IONM arm

SUMMARY:
Scientific objectives:

Primary objective:

• To assess if the use of IONM can decrease the rates of temporary RLN palsy after thyroid cancer surgery

Secondary objectives:

* To assess if the use of IONM can decrease permanent RLN palsy rates in patients with thyroid cancers
* To assess voice parameters in patients with RLN palsy

Methodology:

All patients undergoing total thyroidectomy with or without central compartment neck dissection, for thyroid cancers, will be eligible for participation. After confirmation of eligibility and obtaining informed consent, all patients will undergo preoperative screening procedures. Fibreoptic laryngoscopy (FOL) examination will be done to document function of the vocal cords. Preoperative voiceevaluation, GRBAS voice scale assessment and Voice Related Quality of Life (VR-QOL) assessment will be performed for all patients. Patients will then be randomized in a 1:1 ratio to receive IONM or not during surgery. Patients will be stratified as per predefined stratification factors. After surgery, endpoint assessment of vocal cord mobility will be done with a FOL study, by an assessor blinded to the randomization arm. Voice evaluation, GRBAS scale assessment and VR QOL assessment will also be done. An event will be defined as any vocal fold paresis/palsy. Patients without the event will be followed up for 6 months while patients with the event will be followed up for 2 years to assess recovery of vocal cord function and changes in speech parameters. All patients with vocal cord paresis/palsy will be given speech and swallowing rehabilitation

DETAILED DESCRIPTION:
Background and rationale of the study:

The incidence of the thyroid carcinoma has dramatically increased in the last few decades.1Total thyroidectomy with or without central compartment dissection is the treatment of choice for thyroid carcinoma. Vocal cord palsy (VCP) due to injury to the recurrent laryngeal nerve (RLN) is one of the most dreaded complications of this surgery. The symptoms associated with this complication include hoarseness of voice, voice fatigue and aspiration. Vocal cord palsy can be either temporary or permanent. The reported incidence of temporary VCP varies from 0-12%.2-4 However, the incidence of permanent VCP has been reported to be much lower varying from 0 to 3.5%.4,5Many patients may not present with symptoms of hoarseness and a post-operative laryngoscopic examination is required in all patients who have undergone surgery for thyroid cancer.6 However, the morbidity associated with VCP significantly affects the quality of life of the patient and at times require intervention to prevent aspiration or to improve voice quality.7 In a recent publication from our institute the invesigator found a temporary VCP rate of 11.8%.8

Intra operative nerve monitoring (IONM) is a technique of monitoring the RLN during surgery, to help identification and safe guarding of the nerve during total thyroidectomy as well as central compartment clearance (CCC). This is a well established technique with many centers in the world routinely using monitoring during surgery. There have been 4 RCTs and 2 meta analysis looking at the role of IONM in decreasing RLN palsy after thyroidectomy. The results from the same have been equivocal with 3 of 4 RCTs showing no added benefit in decreasing RLN palsy rates with the use of IONM.9-12 Of the 2 meta analysis, there was a decrease in RLN palsy rates in one of the meta analysis. 13 however the other Meta analysis by Higgins et al showed no improvement in RLN palsy rates with the use of IONM.14 In the meta analysis by Yang et al, published in 2016, there was a 44% (p=ns) decrease in temporary RLN palsy rates in the thyroid cancer cohort. However, the literature on use of IONM is still equivocal in literature. The other issue with available literature on use of IONM is that, most studies have looked at a heterogenous population of patients being operated for benign and malignant disease. Also most patients in the series evaluated have been patients who have undergone surgery for benign multinodular goiters. The extent of RLN dissection in these patients is limited as compared to patients undergoing surgery for thyroid cancers which involve total thyroidectomy and central compartment dissections. There have been no RCTs looking at the role of IONM in preventing RLN palsy in thyroid cancer surgeries. Also none of the RCTs performed have had a formal sample size calculation and robust analysis.

Section B: Aims and Objectives Aim: To assess the role of IONM in thyroid cancer surgery

Primary objective:

• To assess if the use of IONM can decrease the rates of temporary RLN palsy after thyroid cancer surgery

Secondary objectives:

* To assess if the use of IONM can decrease permanent RLN palsy rates in patients with thyroid cancers
* To assess voice parameters in patients with RLN palsy

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy with or without central compartment dissection
* Redo total/completion thyroidectomy

Exclusion Criteria:

* Patients operated for benign diseases
* Hemithyroidectomy
* Pre operative cord fixity
* High risk for intraoperative RLN sacrifice as determined by the treating surgeon
* Redo patients undergoing unilateral procedures
* Patients unwilling to participate in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Primary objective assessment (Temporary RLN palsy)- FOL evaluation | upto 21 days after surgery
  The vocal cord mobility of each patient will be documented as mobile, fixed or restricted. Restriction of VC movement will be considered as an event for analysis. Other parameters like phonatory gap, arytenoid position, aspiration evaluation will also be done and recorded.

SECONDARY OUTCOMES:
Acoustic analysis | upto 21 days
  Dr Speech software
Aerodynamic voice measurement | upto 21 days after surgery
  Maximum Phonation time
Voice quality assessment | upto 21 days after surgery
  GRBAS score (Grade of Roughness, Breathiness, Asthenia and Strain)

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Parel, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
Yes